CLINICAL TRIAL: NCT01558232
Title: A Prospective, Experimental ABA Study to Evaluate Use of the Tibion Bionic Leg in Subacute Post-stroke Patients Undergoing Physical Therapy
Brief Title: A Prospective Study to Evaluate Use of the Tibion Bionic Leg in Sub-Acute Post-stroke Patients
Acronym: Acute Effects
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was terminated base on Sponsor's decision.
Sponsor: Tibion Bionics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP001
Record Dates: First submitted 2012-03-06; First posted 2012-03-20 (Estimated); Last update posted 2012-07-09 (Estimated); Status verified 2012-07

CONDITIONS: Stroke
Keywords: Stroke; Tibion; Bionics; Rehab; Therapy; Robotics; Intention
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tibion Arm (Experimental): Arm of the study in which enrolled subacute post-stroke subjects undergo lower extremity physical therapy using the Tibion Bionic Leg.
  Interventions: Device: Tibion Bionic Leg

INTERVENTIONS:
Device: Tibion Bionic Leg — The Tibion Bionic Leg is used as an adjunct in post-stroke and post-operative rehabilitative physical therapy. The leg is a lightweight, wearable, portable, battery-powered, motorized leg orthosis that provides active assistance and resistance to lower limb movement during walking, stair ascent and descent, and transfers from sitting to standing (and standing to sitting).

SUMMARY:
The objective of this clinical study is to examine acute changes in stability, force allocation, work, and mobility from using a wearable, portable, battery-operated robotic orthosis (the Tibion Bionic Leg) in subacute post-stroke persons undergoing lower extremity physical therapy.

DETAILED DESCRIPTION:
Samples text.

ELIGIBILITY:
Inclusion Criteria:

* Single stroke with residual unilateral lower-extremity weakness
* Subacute post-stroke period (>3 and <12 months)
* Eligible to participate to lower extremity physical therapy
* Age 40 years or greater
* Able to ambulate at least 10 meters
* Able to ambulate without a leg brace
* Ambulation speed less than 0.8 meters/second
* Minimum to moderate assist for transfer or ambulation by physical therapist evaluation
* Subject must understand the nature of the study and provide written informed consent prior to enrollment.
* Subject must be willing and able to attend all study sessions

Exclusion Criteria:

* Medically unstable
* Age younger than 40 years
* Acute post-stroke (< 3 months)
* Chronic post-stroke (> 12 months)
* Status-post multiple strokes
* Status-post traumatic brain injury
* Ambulation speed greater than 0.8 meters/second
* Currently using a Knee-Ankle-Foot Orthosis (KAFO)
* Not eligible for lower extremity physical therapy
* Concomitant degenerative neurological conditions
* Not able to ambulate at least 10 meters without assistance
* Greater than moderate assist during transfer or ambulation by physical therapist evaluation
* Unable to ambulate without a leg brace
* Unable to follow instructions, complete follow-up, or provide informed consent.
* Currently enrolled in another investigational device or drug trial

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2012-03; Primary Completion 2012-08 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Ambulation Speed | Baseline (prior to training); at conclusion of training regimen, an average of 2 weeks.
  Walking speed (comfortable and fastest possible), in meters per second, as measured by the 10 Meter Walk Test (10 MWT).

SECONDARY OUTCOMES:
Measurements of Gait | Baseline (prior to training); prior to the first training session; prior to the second training session; at the conclusion of training regimen completed an average of 2 weeks.
  The secondary endpoints are obtained from the GAITRite analysis system:
  * Measurements of gait, such as the length and time of step, cycle, and stride, Heel to Heel base support, single/double limb support time, and stance and swing phase timing.
Measurements of Stride | Baseline (prior to training); prior to the first training session; prior to the second training session; at the conclusion of training regimen completed an average of 2 weeks.
  Other secondary endpoints are obtained from the GAITRite analysis system:
  * Measurements of Stride such as distance, ambulation time, velocity, normalized velocity, cadence, step time, step length, cycle time.
Measurements of Force, Stance, and Stability | Baseline (prior to training); prior to the first training session; prior to the second training session; at the conclusion of training regimen completed an average of 2 weeks.
  Other secondary endpoints are obtained from Balance Master system:
  * Limb parameters, including force in transfers from sitting to standing, standing to sitting, weight-bearing squats, and limits of stability.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Browne, MD, Principal Investigator — Magee Rehabilitation Hospital
Locations (1):
- Magee Rehabilitation Hospital, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Wong CK, Bishop L, Stein J. A wearable robotic knee orthosis for gait training: a case-series of hemiparetic stroke survivors. Prosthet Orthot Int. 2012 Mar;36(1):113-20. doi: 10.1177/0309364611428235. Epub 2011 Nov 14. PMID 22082495
- [Background] Horst RW. A bio-robotic leg orthosis for rehabilitation and mobility enhancement. Annu Int Conf IEEE Eng Med Biol Soc. 2009;2009:5030-3. doi: 10.1109/IEMBS.2009.5333581. PMID 19964374
- [Background] Horst RW, Marcus RR. FlexCVA: a continuously variable actuator for active orthotics. Conf Proc IEEE Eng Med Biol Soc. 2006;2006:2425-8. doi: 10.1109/IEMBS.2006.259950. PMID 17946511
- See also: Tibion Bionic Leg — http://www.tibion.com